CLINICAL TRIAL: NCT04142008
Title: Walk With Me: a Mobile Application to Improve Walking in Persons With MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Peter Feys, Principal Investigator, Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: B9115201836734
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Walk with Me app (Experimental)
  Interventions: Device: Walk with Me app

INTERVENTIONS:
Device: Walk with Me app — For 10 weeks the subjects will use a mobile application (Walk with Me). The aim of this study is to investigate the usability of the mobile application, as well as investigating if the mobile application effects walking

SUMMARY:
During 10 weeks the subjects will use a mobile application (Walk with Me). The aim of this study is to investigate the usability of the mobile application, as well as investigating if the mobile application effects walking.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis according to the McDonald Criteria
* Able to walk independently or with unilateral support for 10 minutes

Exclusion Criteria:

* Exacerbation or relapse within last 3 months before study
* Other medical condition interfering with walking ability (e.g. cardiac or respiratory diseases, arthritis and fibromyalgia, stroke, Parkinson).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
VAS score pre 6-minute walk test (6 MWT) indoor | Baseline
  he instructor will ask the participant to rate their fatigue from 0-10 (0= no fatigue, 10= most fatigued ever)
VAS score pre 6-minute walk test (6 MWT) outdoor | Baseline
  he instructor will ask the participant to rate their fatigue from 0-10 (0= no fatigue, 10= most fatigued ever)
VAS score pre 6-minute walk test (6 MWT) indoor | week 11
  he instructor will ask the participant to rate their fatigue from 0-10 (0= no fatigue, 10= most fatigued ever)
VAS score pre 6-minute walk test (6 MWT) outdoor | Baseline
  Participants will be instructed to perform the 6MWT. After this test the instructor will ask the participant to rate their fatigue from 0-10 (0= no fatigue, 10= most fatigued ever).
VAS score pre 6-minute walk test (6 MWT) indoor | week 11
  Participants will be instructed to perform the 6MWT. After this test the instructor will ask the participant to rate their fatigue from 0-10 (0= no fatigue, 10= most fatigued ever).
VAS score pre 6-minute walk test (6 MWT) outdoor | week 11
  Participants will be instructed to perform the 6MWT. After this test the instructor will ask the participant to rate their fatigue from 0-10 (0= no fatigue, 10= most fatigued ever).
Distance walked index during the 6MWT indoor | Baseline
  During this test participants are instructed to walk as far as possible on a 30-meter course for 6 minutes. The distance walked is recorded every minute. The distance of the last minute is compared to the distance walked in the first minute to find the index.
Distance walked index during the 6MWT outdoor | Baseline
  During this test participants are instructed to walk as far as possible on a 30-meter course for 6 minutes. The distance walked is recorded every minute. The distance of the last minute is compared to the distance walked in the first minute to find the index.
Distance walked index during the 6MWT indoor | week 11
  During this test participants are instructed to walk as far as possible on a 30-meter course for 6 minutes. The distance walked is recorded every minute. The distance of the last minute is compared to the distance walked in the first minute to find the index.
Distance walked index during the 6MWT outdoor | week 11
  During this test participants are instructed to walk as far as possible on a 30-meter course for 6 minutes. The distance walked is recorded every minute. The distance of the last minute is compared to the distance walked in the first minute to find the index.
MSWS-12 score | Baseline
  This is a short questionnaire to map out walking difficulties in daily living.
MSWS-12 score | Week 11
  This is a short questionnaire to map out walking difficulties in daily living.
the Paced Auditory Serial Addition Test (PASAT) (Cognitive Fatigability) | baseline
  This is a cognitive test where the participant will try to retain certain numbers they hear and do math. Correct answer last 1/3 vs first 1/3
the Paced Auditory Serial Addition Test (PASAT) (Cognitive Fatigability) | week 11
  This is a cognitive test where the participant will try to retain certain numbers they hear and do math. Correct answer last 1/3 vs first 1/3
the Symbol Digit Modality Test (SDMT) (Cognitive fatigability) | baseline
  his is a cognitive performance test, substantiated with focus, speed, and visual scanning. Correct answers last 30 seconds vs first 30 seconds
the Symbol Digit Modality Test (SDMT) (Cognitive fatigability) | week 11
  his is a cognitive performance test, substantiated with focus, speed, and visual scanning. Correct answers last 30 seconds vs first 30 seconds

SECONDARY OUTCOMES:
5 times sit to stand (5xSTS) (Motor Function test) | Baseline
  This is a motor test to assess the functional lower limb muscle strength. The participant is asked to stand from a seated position and sit down again as fast as possible for five times in a row.
5 times sit to stand (5xSTS) (Motor Function test) | Week 11
  This is a motor test to assess the functional lower limb muscle strength. The participant is asked to stand from a seated position and sit down again as fast as possible for five times in a row.
Timed 25 Foot Walk (T25FW) (Motor Function) | baseline
  This is a motor test at which the participant is instructed to walk 25 ft (=7,62 meter) as fast and safely as possible. This is a quantitative performance test to assess mobility and leg function.
Timed 25 Foot Walk (T25FW) (Motor Function) | week 11
  This is a motor test at which the participant is instructed to walk 25 ft (=7,62 meter) as fast and safely as possible. This is a quantitative performance test to assess mobility and leg function.
Nine Hole Peg Test (NHPT) | baseline
  This is a motor test to assess the participant's manual skills. This test records the time the participant needs to place 9 pins in the pegboard and remove them again.
Nine Hole Peg Test (NHPT) | week 11
  This is a motor test to assess the participant's manual skills. This test records the time the participant needs to place 9 pins in the pegboard and remove them again.
Modified Fatigue Impact Scale (MFIS) | baseline
  This is a short questionnaire to evaluate to impact of general fatigue. This questionnaire measures the effects of fatigue on three levels: physical, cognitive and psychosocial.
Modified Fatigue Impact Scale (MFIS) | Week 11
  This is a short questionnaire to evaluate to impact of general fatigue. This questionnaire measures the effects of fatigue on three levels: physical, cognitive and psychosocial.
Fatigue severity scale (FSS) | baseline
  This is a short questionnaire to measure the severity of general fatigue.
Fatigue severity scale (FSS) | week 11
  This is a short questionnaire to measure the severity of general fatigue.
Multiple Sclerosis Impact Scale (MSIS-29) | baseline
  This is a short self-report questionnaire used to assess the day-to-day life in the past two weeks. This questionnaire has a physical and psychological scale.
Multiple Sclerosis Impact Scale (MSIS-29) | week 11
  This is a short self-report questionnaire used to assess the day-to-day life in the past two weeks. This questionnaire has a physical and psychological scale.
Health-related quality of life (SF-36) | baseline
  This is a short questionnaire to measure health status.
Health-related quality of life (SF-36) | week 11
  This is a short questionnaire to measure health status.
International Physical Activity Questionnaire (IPAQ) | baseline
  This is a questionnaire to measure health-related physical activity
International Physical Activity Questionnaire (IPAQ) | week 11
  This is a questionnaire to measure health-related physical activity

CONTACTS AND LOCATIONS:
Overall Officials: peter Feys, prof. dr., Principal Investigator — Hasselt University; Fanny Van Geel, drs., Study Chair — Hasselt University
Locations (1):
- Hasselt University, Hasselt, Belgium